CLINICAL TRIAL: NCT03739996
Title: A Study of Long-Acting Cabotegravir Plus VRC-HIVMAB075-00-AB (VRC07-523LS) to Maintain Viral Suppression in Adults Living With HIV-1
Brief Title: Long-Acting Cabotegravir Plus VRC-HIVMAB075-00-AB (VRC07-523LS) for Viral Suppression in Adults Living With HIV-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5357; 30005 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CAB LA + VRC07-523LS (Experimental): Step 1: CAB administered orally as one 30 mg tablet once daily, plus two NRTIs, for up to 5 weeks.
  Step 2: CAB LA loading dose (600 mg) administered as one IM injection at Step 2 entry study visit, and maintenance dose (400 mg), starting at 4 weeks after CAB LA loading dose, and then every 4 weeks through Week R2+44 (for a total of 12 injections).
  VRC07-523LS (40 mg/kg) administered as an IV infusion starting at Step 2 entry and then every 8 weeks through Week R2+40 (for a total of 6 infusions).
  Step 3: Standard of Care (SOC) ART regimen for approximately 48 weeks.
  Interventions: Drug: Oral Cabotegravir (CAB); Drug: Nucleoside Reverse Transcriptase Inhibitors (NRTIs); Drug: Long-Acting Injectable Cabotegravir (CAB LA); Biological: VRC07-523LS; Drug: Standard of Care (SOC) ART

INTERVENTIONS:
Drug: Oral Cabotegravir (CAB) — 30 mg tablets administered orally
Drug: Nucleoside Reverse Transcriptase Inhibitors (NRTIs) — NRTIs were not provided by the study. Participants obtained NRTIs outside of the study through routine care.
Drug: Long-Acting Injectable Cabotegravir (CAB LA) — 600 mg loading dose followed by 400 mg maintenance doses administered by intramuscular (IM) injection
Biological: VRC07-523LS — 40 mg/kg administered as an intravenous (IV) infusion
  Other Names: VRC-HIVMAB075-00-AB
Drug: Standard of Care (SOC) ART — SOC ART was not provided by the study. Participants obtained SOC ART outside of the study through routine care.

SUMMARY:
The purpose of this study was to assess the safety, tolerability, antiviral activity, and pharmacokinetics of long-acting cabotegravir (CAB LA) plus the broadly neutralizing monoclonal antibody VRC-HIVMAB075-00-AB (VRC07-523LS), in adults living with HIV-1 with suppressed plasma viremia.

DETAILED DESCRIPTION:
This study had a single, open-label arm and was conducted in three steps.

At Step 1 entry, all participants discontinued their current antiretroviral therapy (ART) regimen, except for the 2 nucleoside reverse transcriptase inhibitors (NRTIs) and started oral CAB. Viral load monitoring occurred at entry, Week 4, and, conditionally, Week 5.

During Step 1, participants who tolerated oral CAB plus their two NRTIs, maintained viral suppression, and met the other Step 2 eligibility requirements, registered for Step 2. Participants in Step 1 who were not eligible for Step 2 returned to their standard of care (SOC) regimen and were followed for an additional 4 weeks before being taken off the study.

In Step 2, participants received CAB LA every 4 weeks through Step 2 Week 44 (12 injections) plus VRC07-523LS every 8 weeks through Step 2 Week 40 (6 infusions). Viral load monitoring occurred every 2 weeks through Week 8 and then every 4 weeks through Week 48. Any participant with a viral load of HIV-1 RNA ≥ 200 copies/mL had to attend an additional virologic failure confirmation visit within 14 days of the measured value. If virologic failure was confirmed (i.e., two consecutive HIV-1 RNA values ≥ 200 copies/mL), the participant transitioned to Step 3.

After completion of Step 2 (Week 48), confirmed virologic failure, or premature treatment discontinuation, all participants who received any CAB LA or VRC07-523LS entered Step 3 and returned to SOC ART for 48 weeks, with visits at step entry and weeks 4, 12, 24, 36, and 48.

The study's primary virology outcome pertains to Step 2 and only includes participants who started the CAB LA plus VRC07-523LS combination. The study's primary safety outcome pertains to Step 2 and Step 3 follow-up for participants who started the CAB LA plus VRC07-523LS combination.

Study visits included physical examinations, clinical assessments, and blood and urine collection.

The study opened to accrual in late December 2019. However, in March 2020 the study temporarily closed to screening and enrollment (including registration to Step 2) due to the COVID-19 pandemic. No participant had reached Step 2 of the study when the pause occurred. Participants in Step 1 were instructed to immediately stop the oral CAB plus 2 NRTI combination, resume their SOC regimen, and discontinue the study. The study reopened to screening and enrollment in September 2020. Analyses for this study only included participants who enrolled after the study reopened in September 2020. Participants previously enrolled were invited to rescreen and reenroll, if still eligible.

ELIGIBILITY:
Step 1 Inclusion Criteria:

* Individual with HIV-1
* On a three-drug ART regimen for at least 8 weeks that includes a boosted protease inhibitor (PI), a nonnuceloside reverse transcriptase inhibitor (NNRTI), or an integrase inhibitor (INSTI) plus two nuclesodie reverse transcriptase inhibitors (NRTI) with no history of switch due to virologic failure.
* CD4+ cell count greater than or equal to 350 cells/mm^3
* Virally suppressed (< 50 copies/mL) within 2 years prior to study entry
* Susceptibility to VRC07-523LS based on IC50 less than or equal to 0.25 ug/mL and a Maximum Percent Inhibition > 98% using the Monogram PhenoSense Assay
* Certain laboratory values obtained within 60 days prior to study entry and in an acceptable range
* For participants of child-bearing potential:

  * A negative serum or urine pregnancy test within 48 hours prior to study entry
  * If participating in sexual activity that could lead to pregnancy, must agree to use an effective form of contraception.
* Negative HBsAg result
* Negative hepatitis C virus antibody
* Ability and willingness to provide written informed consent

Step 1 Exclusion Criteria:

* Any previous receipt of humanized or human monoclonal antibody (licensed or investigational).
* Weight greater than 115 kg or less than 53 kg.
* AIDS-defining illness within 60 days prior to study entry.
* History of a severe allergic reaction within 2 years prior to study entry.
* Currently breastfeeding or pregnant.
* Active drug or alcohol use or dependence that would interfere with adherence to study requirements.
* Acute or serious illness that requires systemic treatment, quarantine, and/or hospitalization within 30 days prior to entry.
* Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 60 days prior to study entry.
* Treatment for hepatitis C within 24 weeks prior to study entry.
* Vaccinations within 7 days prior to study entry.
* Initiation of ART during acute HIV-1 infection (as determined by the site investigator by history and/or available medical records).
* Personal or known family history of prolonged QT syndrome or a clinically significant finding on the screening electrocardiogram (ECG) based on an assessment of the screening ECG by that site investigator.
* Unstable liver disease or known biliary abnormalities
* Moderate or severe hepatic impairment (Class B or C) as determined by Child-Pugh classification.
* History of seizures or treatment for seizures within the past 2 years prior to study entry.
* Current acute illness that in the opinion of the investigator will prevent the participant from complying with study visits.

Step 2 Inclusion Criteria:

* HIV-1 RNA less than 50 copies/mL at week 4 (Step 1), or HIV-1 RNA of 50-199 copies/mL at week 4 followed by HIV-1 RNA less than 50 copies/mL at week 5 (Step 1).
* For participants of child-bearing potential:

  * A negative serum or urine pregnancy test within 48 hours prior to step 2 entry
  * If participating in sexual activity that could lead to pregnancy, continued agreement to use an effective form of contraception.

Step 2 Exclusion Criteria:

* Discontinuation or temporary hold of oral CAB or NRTIs for greater than 7 consecutive days for any reason during Step 1.
* Grade 3 or 4 adverse event thought to be related to oral CAB during Step 1 according to the site investigator.
* Vaccination (e.g., influenza) within 7 days prior to the Step 2 registration.
* Currently breastfeeding or pregnant.
* Any greater than or equal to Grade 2 ALT (greater than 2.5 times ULN) that developed during Step 1.

Step 3 Inclusion Criterion:

* Received any CAB LA or VRC07-523LS during Step 2.

Step 3 Exclusion Criterion:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-12-31 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Babafemi Taiwo, MBBS, Study Chair — Northwestern University CRS; Pablo Tebas, MD, Study Chair — Hospital of the University of Pennsylvania CRS; Leah Burke, MD, Study Chair — Weill Cornell Chelsea CRS
Locations (18):
- United States (17):
  - Alabama CRS, Birmingham, Alabama
  - UCSD Antiviral Research Center CRS, San Diego, California
  - Ucsf Hiv/Aids Crs, San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Northwestern University CRS, Chicago, Illinois
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - Weill Cornell Chelsea CRS, New York, New York
  - Columbia P&S CRS, New York, New York
  - Weill Cornell Uptown CRS, New York, New York
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS, Rochester, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Cincinnati Clinical Research Site, Cincinnati, Ohio
  - Ohio State University CRS, Columbus, Ohio
  - Penn Therapeutics, CRS, Philadelphia, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico AIDS Clinical Trials Unit CRS, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the Advancing Clinical Therapeutics Globally (ACTG) by NIH.
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the ACTG.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the ACTG.
  * By what mechanism will data be made available?
    * Researchers may submit a request for access to data using the ACTG "Data Request" form at:https://submit.mis.s-3.net/ Researchers of approved proposals will need to sign an ACTG Data Use Agreement before receiving the data.

REFERENCES:
- [Derived] Kuritzkes DR. Broadly neutralizing antibodies and long-acting antiretroviral drugs as treatments for HIV. Curr Opin HIV AIDS. 2023 Jul 1;18(4):225-228. doi: 10.1097/COH.0000000000000801. Epub 2023 May 9. PMID 37265259
- See also: The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017 — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled from Dec 2019 to May 2022 at 18 sites in the United States. In Mar 2020 the study temporarily closed to screening and enrollment. During this pause, all participants were taken off the study. The study reopened to screening and enrollment in mid-September 2020. Analyses only included participants who enrolled after the study reopened. All previously enrolled participants were encouraged to return and rescreen.
  Note: Not all participants who entered Step 1, entered Step 2.
Pre-assignment Details: There was no randomization in this study.
Groups:
- CAB LA + VRC07-523LS: Step 1: CAB administered orally as one 30 mg tablet once daily, plus two NRTIs, for up to 5 weeks.
  Step 2: CAB LA loading dose (600 mg) administered as one IM injection at Step 2 entry study visit, and maintenance dose (400 mg), starting at 4 weeks after CAB LA loading dose, and then every 4 weeks through Week R2+44 (for a total of 12 injections).
  VRC07-523LS (40 mg/kg) administered as an IV infusion starting at Step 2 entry and then every 8 weeks through Week R2+40 (for a total of 6 infusions).
  Step 3: Standard of Care (SOC) ART regimen for approximately 48 weeks.
  Oral Cabotegravir (CAB): 30 mg tablets administered orally
  Nucleoside Reverse Transcriptase Inhibitors (NRTIs): NRTIs were not provided by the study. Participants obtained NRTIs outside of the study through routine care.
  Long-Acting Injectable Cabotegravir (CAB LA): 600 mg loading dose followed by 400 mg maintenance doses administered by intramuscular (IM) injection
  VRC07-523LS: 40 mg/kg administered as an intravenous (IV) infusion
  Standard of Care (SOC) ART: SOC ART was not provided by the study. Participants obtained SOC ART outside of the study through routine care.
Period: Step 1 (Oral CAB + 2 NRTIs)
Arm/Group | CAB LA + VRC07-523LS
Started | 75
Completed Step 1 and Enrolled to Step 2 | 71
Completed Step 1 and Discontinued the Study | 3
Completed | 74
Not Completed | 1
Not completed — Determined to be ineligible | 1
Period: Step 2 (CAB LA + VRC07-523LS)
Arm/Group | CAB LA + VRC07-523LS
Started | 71 (Not all participants who completed Step 1 treatment moved on to Step 2.)
Completed Step 2 and Enrolled to Step 3 | 60
Prematurely Discontinued Step 2 and Enrolled to Step 3 | 8
Prematurely Discontinued Step 2 and Discontinued the Study | 3
Completed | 60 (Participants did not have to complete Step 2 to advance to Step 3. All participants who received any dose of CAB LA or VRC07-523LS in Step 2 registered to Step 3 at the final Step 2 visit, at confirmed virologic failure, or at premature treatment discontinuation.)
Not Completed | 11
Not completed — Death | 1
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Virologic failure, as defined by the protocol | 5
Not completed — Participant refusal to remain on long-acting treatment | 3
Period: Step 3 (SOC ART)
Arm/Group | CAB LA + VRC07-523LS
Started | 68 (Participants did not have to complete Step 2 to advance to Step 3. All participants who received any dose of CAB LA or VRC07-523LS in Step 2 registered to Step 3 at the final Step 2 visit, at confirmed virologic failure, or at premature treatment discontinuation.)
Completed | 66
Not Completed | 2
Not completed — Death | 1
Not completed — Participant moved | 1

BASELINE CHARACTERISTICS:
Population: 75 participants were enrolled to the study. One participant enrolled erroneously despite not meeting the eligibility criteria for VRC07-523LS susceptibility. This participant discontinued the study during Step 1 and is excluded from all analyses.
Arm/Group | CAB LA + VRC07-523LS
Number analyzed (Participants) | 74
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [46 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White (Non-Hispanic) | 38
  Black (Non-Hispanic) | 25
  Hispanic or Latino (regardless of race) | 8
  Other | 3
Baseline BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 28 [25 to 32]
Baseline HIV-1 RNA [Count of Participants; unit: Participants]
  Less than 50 copies/mL | 71
  Greater than or equal to 50 copies/mL | 3
Baseline CD4 cell count [Median (Inter-Quartile Range); unit: cells/mm^3] — Population: One participant had a missing CD4 count at study entry.
  cells/mm^3
    number analyzed (Participants) | 73
    (all) | 720 [570 to 895]
VRC07-523LS IC50 [Median (Full Range); unit: ug/mL] — The IC50 represents the VRC07-523LS concentration needed to inhibit viral replication by 50%.
  ug/mL | 0.076 [0.019 to 0.249]
VRC07-523LS MPI [Median (Full Range); unit: Percent] — The Maximum Percent Inhibition (MPI) refers to the highest level of viral replication inhibition achieved by a specific VRC07-523LS concentration.
  Percent | 99.9 [98.5 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Experiencing a Grade 3 or Higher Adverse Event (AE) or Premature Discontinuation Due to an AE (Regardless of Grade) That is Related To Step 2 Study Treatment (CAB LA Plus VRC07-523LS)
Description: The proportion of participants reporting a grade 3 (severe), grade 4 (potentially life-threatening), or grade 5 (death) adverse event OR premature discontinuation due to an adverse event (regardless of grade) that the clinical management committee judged to be at least possibly related to the CAB LA plus VRC07-523LS combination.
  Based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017
Time Frame: Measured from Step 2 entry through the remaining study follow-up (e.g., any time on Step 2 or Step 3 for a maximum follow-up time of 96 weeks).
Population: All participants who initiated the CAB LA plus VRC07-523LS combination
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | CAB LA + VRC07-523LS
Number analyzed (Participants) | 71
Proportion of participants | 0.17 [0.10 to 0.27]

2. Primary Outcome: Cumulative Probability of Confirmed Virologic Failure at or Prior to Step 2 Week 44
Description: Virologic failure is defined as confirmed (i.e., two consecutive values) HIV-1 RNA ≥ 200 copies/mL at or prior to Step 2 Week 44 of the CAB LA plus VRC07-523LS combination.
Time Frame: Measured from Step 2 entry through Step 2 Week 44
Population: All participants who initiated the CAB LA plus VRC07-523LS combination
Measure: Number (95% Confidence Interval); unit: Cumulative probability
Arm/Group | CAB LA + VRC07-523LS
Number analyzed (Participants) | 71
Cumulative probability | 0.07 [0.03 to 0.16]

3. Secondary Outcome: Median Concentrations of VRC07-523LS
Description: Concentrations of VRC07-523LS, measured in serum, at selected time points in Step 2.
Time Frame: Measured at Step 2 Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48
Population: All participants who initiated the CAB LA plus VRC07-523LS combination and had PK samples obtained at the scheduled study visits were included.
Measure: Median (Inter-Quartile Range); unit: ug/mL
Arm/Group | CAB LA + VRC07-523LS
Number analyzed (Participants) | 69
ug/mL
  Step 2 Week 4: number analyzed (Participants) | 67
  Step 2 Week 4 | 177 [159 to 200]
  Step 2 Week 8 | 105 [92.2 to 121]
  Step 2 Week 12: number analyzed (Participants) | 66
  Step 2 Week 12 | 232 [198 to 279]
  Step 2 Week 16: number analyzed (Participants) | 67
  Step 2 Week 16 | 146 [114 to 160]
  Step 2 Week 20: number analyzed (Participants) | 64
  Step 2 Week 20 | 261 [218 to 297]
  Step 2 Week 24: number analyzed (Participants) | 60
  Step 2 Week 24 | 151 [121 to 174]
  Step 2 Week 28: number analyzed (Participants) | 61
  Step 2 Week 28 | 264 [233 to 306]
  Step 2 Week 32: number analyzed (Participants) | 62
  Step 2 Week 32 | 161 [138 to 185]
  Step 2 Week 36: number analyzed (Participants) | 62
  Step 2 Week 36 | 269 [240 to 297]
  Step 2 Week 40: number analyzed (Participants) | 61
  Step 2 Week 40 | 156 [139 to 185]
  Step 2 Week 44: number analyzed (Participants) | 61
  Step 2 Week 44 | 266 [226 to 306]
  Step 2 Week 48: number analyzed (Participants) | 59
  Step 2 Week 48 | 166 [145 to 190]

4. Secondary Outcome: Median Concentration of CAB LA
Description: Concentrations of long-acting cabotegravir, measured in plasma, at select time points in Step 2
Time Frame: Measured at Step 2 Week 4, 8, 24, and 48
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | CAB LA + VRC07-523LS
Number analyzed (Participants) | 70
ng/mL
  Step 2 Week 4: number analyzed (Participants) | 69
  Step 2 Week 4 | 1398 [891 to 2201]
  Step 2 Week 8 | 1714 [1376 to 2503]
  Step 2 Week 24: number analyzed (Participants) | 63
  Step 2 Week 24 | 2386 [1857 to 2886]
  Step 2 Week 48: number analyzed (Participants) | 60
  Step 2 Week 48 | 2760 [2125 to 3234]

5. Secondary Outcome: ARV Resistance of Breakthrough Isolates
Description: ARV resistance testing was conducted on samples obtained when confirmed virologic failure (two consecutive HIV-1 RNA values ≥ 200 copies/mL) occurred. Interpretation of resistance results, pertaining to integrase inhibitor resistance mutations, was obtained using the Stanford HIVDB Algorithm Version 9.3 (released 2022-11-20).
Time Frame: Measured from Step 2 entry through Step 2 Week 48
Population: Participants with confirmed virologic failure (two consecutive HIV-1 RNA values ≥ 200 copies/mL) who initiated the VRC07-523LS + CAB LA combination and had reportable assay results.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + VRC07-523LS
Number analyzed (Participants) | 4
Participants
  Susceptible | 3
  Intermediate or Low-Level Resistance | 1

6. Secondary Outcome: Cumulative Probability of Confirmed Virologic Failure at or Prior to Step 2 Week 24
Description: Virologic failure defined as confirmed (i.e., two consecutive values) HIV-1 RNA ≥ 200 copies/mL
Time Frame: Measured from Step 2 entry through Step 2 Week 24
Population: All participants who initiated the CAB LA plus VRC07-523LS combination
Measure: Number (95% Confidence Interval); unit: Cumulative probability
Arm/Group | CAB LA + VRC07-523LS
Number analyzed (Participants) | 71
Cumulative probability | 0.04 [0.01 to 0.12]

7. Secondary Outcome: Cumulative Probability of Confirmed Virologic Failure or Premature Treatment Discontinuation at or Prior to Step 2 Week 44
Description: Virologic failure, defined as confirmed (i.e., two consecutive values) HIV-1 RNA ≥ 200 copies/mL or premature treatment discontinuation, defined as the date at which a participant ended Step 2 treatment (CAB LA and VRC07-523LS), for any reason, without receiving all 12 CAB LA injections and 6 VRC07-523LS infusions, at or prior to Step 2 Week 44.
Time Frame: Measured from Step 2 entry through Step 2 Week 44
Population: All participants initiating the CAB LA plus VRC07-523LS combination
Measure: Number (95% Confidence Interval); unit: Cumulative probability
Arm/Group | CAB LA + VRC07-523LS
Number analyzed (Participants) | 71
Cumulative probability | 0.14 [0.08 to 0.24]

8. Secondary Outcome: Cumulative Probability of Confirmed HIV-1 RNA ≥ 50 Copies/mL at or Prior to Step 2 Week 44
Description: Confirmed (i.e., two consecutive values) HIV-1 RNA ≥ 50 copies/mL measured at or prior to Step 2 Week 44.
Time Frame: Measured from Step 2 entry through Step 2 Week 44
Population: All participants who intiated the CAB LA plus VRC07-523LS combination
Measure: Number (95% Confidence Interval); unit: Cumulative probability
Arm/Group | CAB LA + VRC07-523LS
Number analyzed (Participants) | 71
Cumulative probability | 0.13 [0.07 to 0.23]

9. Secondary Outcome: Cumulative Probability of Confirmed HIV-1 RNA ≥ 50 Copies/mL at or Prior to Step 2 Week 24
Description: Confirmed (i.e., two consecutive values) HIV-1 RNA ≥ 50 copies/mL measured at or prior to Step 2 Week 24.
Time Frame: Measured from Step 2 entry through Step 2 Week 24
Population: All participants who initiated the CAB LA plus VRC07-523LS combination
Measure: Number (95% Confidence Interval); unit: Cumulative probability
Arm/Group | CAB LA + VRC07-523LS
Number analyzed (Participants) | 71
Cumulative probability | 0.12 [0.06 to 0.21]

10. Secondary Outcome: Cumulative Probability of Confirmed HIV-1 RNA ≥ 50 Copies/mL or Premature Treatment Discontinuation at or Prior to Step 2 Week 44
Description: Confirmed (i.e., two consecutive values) HIV-1 RNA ≥ 50 copies/mL or premature treatment discontinuation, defined as the date at which a participant ended Step 2 treatment (CAB LA and VRC07-523LS), for any reason, without receiving all 12 CAB LA injections and 6 VRC07-523LS infusions, at or prior to Step 2 Week 44.
Time Frame: Measured from Step 2 entry through Step 2 Week 44
Population: All participants who initiated the CAB LA plus VRC07-523LS combination
Measure: Number (95% Confidence Interval); unit: Cumulative probability
Arm/Group | CAB LA + VRC07-523LS
Number analyzed (Participants) | 71
Cumulative probability | 0.20 [0.12 to 0.30]

11. Secondary Outcome: Proportion of Participants With HIV-1 RNA ≥ 50 Copies/mL at Step 2 Week 44
Description: The proportion of participants with HIV-1 RNA ≥ 50 copies/mL, HIV-1 RNA < 50 copies/mL, and without data in Step 2 Week 44 window (days 295-322 from Step 2 entry) as defined by the FDA Snapshot algorithm.
Time Frame: Step 2 Week 44
Population: All participants who initiated the CAB LA plus VRC07 combination.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + VRC07-523LS
Number analyzed (Participants) | 71
Participants
  HIV-1 RNA ≥ 50 copies/mL on treatment | 7
  HIV-1 RNA < 50 copies/mL on treatment | 58
  No Virologic Data in Week 44 Window: Disc study/study drug due to an AE or death | 3
  No Virologic Data in Week 44 Window: Disc study/study drug for other reasons | 2
  No Virologic Data in Week 44 Window: On study but missing data in window | 1

12. Secondary Outcome: Frequency of Anti-Drug Antibodies (ADA) Against VRC07-523LS
Description: Number of participants who were anti-drug antibody (ADA) negative or ADA positive calculated at each sampled timepoint.
Time Frame: Measured at Step 2 Week 28 and 48
Population: All participants who initiated the CAB LA plus VRC07-523LS combination and had ADA samples obtained at the scheduled study visit were included.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + VRC07-523LS
Number analyzed (Participants) | 61
Participants
  Step 2 Week 28: ADA Negative | 61
  Step 2 Week 28: ADA Positive | 0
  Step 2 Week 48: number analyzed (Participants) | 59
  Step 2 Week 48: ADA Negative | 59
  Step 2 Week 48: ADA Positive | 0

13. Secondary Outcome: Proportion of Participants Experiencing a Grade 3 or Higher Adverse Event (AE) or Premature Discontinued Due to an AE (Regardless of Grade) That is Related to Oral CAB.
Description: The proportion of participants reporting a grade 3 (severe), grade 4 (potentially life-threatening), or grade 5 (death) adverse event OR premature discontinuation due to an adverse event (regardless of grade) that the clinical management committee judged to be at least possibly related to oral CAB.
  Based on the Division of AIDS Table for Grading the Severity of Adult and Pedatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017.
Time Frame: Measured from Step 1 entry through the end of Step 1 (for a maximum of 5 weeks)
Population: All eligible participants who initiated oral CAB.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | CAB LA + VRC07-523LS
Number analyzed (Participants) | 74
Proportion of participants | 0 [0.0 to 0.05]

14. Secondary Outcome: Proportion of Participants Who Prematurely Discontinued Oral CAB or the CAB LA Plus VRC07-523LS Combination
Description: The proportion of participants who discontinued, for any reason, oral CAB (during Step 1) or the CAB LA plus VRC07-523LS combination.
Time Frame: Measured from Step 1 entry through the end of Step 2 (for a maximum of 53 weeks)
Population: All eligible participants who initiated Step 1 (oral CAB) and all participants who initiated Step 2 (CAB LA plus VRC07-523LS) treatment
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + VRC07-523LS
Number analyzed (Participants) | 74
Participants | 10

15. Secondary Outcome: Proportion of Participants Experiencing a Grade 3 or Higher Adverse Event (AE) That is Related to Oral CAB or the CAB LA Plus VRC07-523LS Combination.
Description: The proportion of participants reporting a grade 3 (severe), grade 4 (potentially life-threatening), or grade 5 (death) that the clinical management committee judged to be at least possibly related to oral CAB or the CAB LA plus VRC07-523LS combination.
  Based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017.
Time Frame: Measured from Step 1 entry through entire study follow-up (for a maximum of 101 weeks)
Population: All eligible participants who initiated oral CAB and all participants who initiated the CAB LA plus VRC07-523LS combination
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | CAB LA + VRC07-523LS
Number analyzed (Participants) | 74
Proportion of participants | 0.15 [.09 to .25]

ADVERSE EVENTS:
Time Frame: Step 1: From study entry through step completion or premature discontinuation of study/Step 1 (maximum time in Step 1 was 5 weeks). Step 2: From Step 2 entry through step completion or premature discontinuation of study/Step 2 (maximum time in Step 2 was 48 weeks). Step 3: From Step 3 entry through study completion of premature discontinuation (maximum time in Step 3 was 48 weeks).
Description: * Grade ≥ 3 AEs
  * Grade ≥ 2 lab findings
  * All AEs that led to a change in study treatment, regardless of grade
  * All AEs meeting SAE definition or EAE reporting requirement
  The DAIDS AE Grading Table (V2.1), July 2017 was used. All eligible participants who entered Step 1 are included. For eligible participants who entered Step 2, AEs occurring in Step 2 are shown separately. All participants in Step 2 were eligible for Step 3. AEs occurring in Step 3 are shown in a separate column.
Groups:
- Step 1: Oral CAB Plus 2 NRTIs: Step 1: CAB administered orally as one 30 mg tablet once daily, plus two NRTIs, for up to 5 weeks.
  Oral Cabotegravir (CAB): 30 mg tablets administered orally Nucleoside Reverse Transcriptase Inhibitors (NRTIs): NRTIs were not provided by the study. Participants obtained NRTIs outside of the study through routine care.
- Step 2: CAB LA + VRC07-523LS: Step 2: CAB LA loading dose (600 mg) administered as one IM injection at Step 2 entry study visit, and maintenance dose (400 mg), starting at 4 weeks after CAB LA loading dose, and then every 4 weeks through Week R2+44 (for a total of 12 injections).
  VRC07-523LS (40 mg/kg) administered as an IV infusion starting at Step 2 entry and then every 8 weeks through Week R2+40 (for a total of 6 infusions).
  Long-Acting Injectable Cabotegravir (CAB LA): 600 mg loading dose followed by 400 mg maintenance doses administered by intramuscular (IM) injection VRC07-523LS: 40 mg/kg administered as an intravenous (IV) infusion
- Step 3: Standard of Care ART: Step 3: Standard of Care (SOC) ART regimen for approximately 48 weeks.
  Standard of Care (SOC) ART: SOC ART was not provided by the study. Participants obtained SOC ART outside of the study through routine care.
Arm/Group | Step 1: Oral CAB Plus 2 NRTIs | Step 2: CAB LA + VRC07-523LS | Step 3: Standard of Care ART
All-Cause Mortality (participants affected / at risk) | 0/74 | 1/71 | 1/68
Serious Adverse Events (participants affected / at risk) | 1/74 | 9/71 | 6/68
Other Adverse Events (participants affected / at risk) | 9/74 | 37/71 | 29/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1: Oral CAB Plus 2 NRTIs (N=74) | Step 2: CAB LA + VRC07-523LS (N=71) | Step 3: Standard of Care ART (N=68)
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 1
Neurosyphilis (Infections and infestations) | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1: Oral CAB Plus 2 NRTIs (N=74) | Step 2: CAB LA + VRC07-523LS (N=71) | Step 3: Standard of Care ART (N=68)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 5 | 0
Fatigue (General disorders) | 0 | 2 | 0
Malaise (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1
Blood bilirubin (Investigations) | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 1
Blood creatine phosphokinase (Investigations) | 0 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 4 | 2
Blood creatinine decreased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 2 | 2
Blood glucose decreased (Investigations) | 0 | 2 | 4
Blood glucose increased (Investigations) | 4 | 4 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0
Creatinine renal clearance decreased (Investigations) | 5 | 14 | 13
Haemoglobin decreased (Investigations) | 0 | 2 | 0
Lipase increased (Investigations) | 2 | 8 | 6
Low density lipoprotein increased (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
Vasospasm (Vascular disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
This single-arm trial was conducted during the COVID-19 and Mpox public health emergencies, which prompted several countermeasures, including widespread use of multiple doses of new vaccines that can potentially impact virologic response.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT03739996/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2023-08-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT03739996/SAP_001.pdf